CLINICAL TRIAL: NCT04948801
Title: SOF/VEL±RBV: Real-World Efficacy and Safety in GT 3 and 6 HCV Patients in China
Brief Title: SOF/VEL±RBV: Efficacy and Safety in GT 3 and 6 HCV Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Zhe-bin Wu, Professor, Third Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: [2018]02-417-01
Record Dates: First submitted 2021-03-16; First posted 2021-07-02 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-07

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — sofosbuvir-velpatasvir drug combination; Sofosbuvir; velpatasvir

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- genotype 3a HCV: genotype 3a hepatitis C
  Interventions: Drug: Epclusa (sofosbuvir and velpatasvir)
- genotype 6 HCV: genotype 6 hepatitis C
  Interventions: Drug: Epclusa (sofosbuvir and velpatasvir)
- genotype 3b HCV: genotype 3b hepatitis C
  Interventions: Drug: Epclusa (sofosbuvir and velpatasvir)

INTERVENTIONS:
Drug: Epclusa (sofosbuvir and velpatasvir) — Epclusa (sofosbuvir and velpatasvir) is a nucleotide analog polymerase inhibitor and pan-genotypic NS5A inhibitor fixed-dose combination for the treatment of chronic genotype 1-6 hepatitis C virus (HCV) infection.

SUMMARY:
150 GT3 or GT6 CHC patients with or without compensated cirrhosis will be recruited from five centers in China including G3a 50, G3b 50, G6 50 respectively. GT3a and GT6 CHC with or without compensated patients will be administered one pill of Epclusa each day for 12 weeks, and GT3b patients will be administered Epclusa each plus Ribavirin for 12 weeks.

DETAILED DESCRIPTION:
This is a Prospective, observational, multi-center, real-world study to investigate real world effectiveness and safety of SOF/VEL±RBV in Chinese patients infected by HCV GT-3 and 6. 150 GT3 or GT6 CHC patients with or without compensated cirrhosis will be recruited from five centers in China including G3a 50, G3b 50, G6 50 respectively. GT3a and GT6 CHC with or without compensated cirrhosis will be administered one pill of Epclusa each day for 12 weeks, and GT3b patients will be administered one pill of Epclusa each plus Ribavirin for 12 weeks.Demographic, clinical, adverse event and virological data were be collected throughout treatment and post-treatment follow-up.

ELIGIBILITY:
Inclusion Criteria:

* HCV RNA ≥ 15 IU/Ml at Screening
* HCV genotype 3a ,3b and 6
* Hepatitis C without decompensated cirrhosis of the liver

Exclusion Criteria:

* Patients failed to previous NS5A-containing DAAs therapy
* Decompensated cirrhosis
* HCC
* Infection with hepatitis B virus (HBV) or human immunodeficiency virus (HIV).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The groups or cohorts will be selected from people who was diagnosed with hepatitis c at the hospital.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-12-08 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
SVR12 | 12 weeks
  HCV RNA <LLOQ at Week 12 after cessation of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Deparment of Infectious Diseases, the Second Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No